CLINICAL TRIAL: NCT00327925
Title: Study to Assess the Effectiveness of the CAAb Test With Ovarian Cancer Patients
Brief Title: Blood Test for Ovarian Cancer Associated Antibodies (CAAb)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lab Discoveries Ltd. (Industry)
Other Study IDs: LD-OC-CAAb
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2006-05

CONDITIONS: Ovarian Cancer
Keywords: Ovarian; Cancer; Antibodies; Ovarian Cancer Associated Antibodies
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Find Cancer Associated Antibodies

SUMMARY:
Blood is collected from patients and cultured in a CimTube (a test tube with stimulation media) for several days. Following the culture step, the supernatant fluid is tested for the presence of CAAb on experimental test kits.

Null Hypothesis: There is no relationship between the presence or absence of ovarian cancer (OC) and the CAAb i.e. d=0.

Alternative Hypothesis: The expectation of the CAAb in the cancer population differs from that of the control population, i.e. m1 is not equal to m2. Since the sign of the difference is not important, the test will be two-sided.

DETAILED DESCRIPTION:
General Information

Antibodies are a specific response to any "foreign" antigen, and they are usually detectable in the serum within 5-7 days after the initial exposure to it. However, there are some cases where there is a suppression of the specific immune response, such as in the case of a tumor. To date, there are no reports on serum antibodies that are associated to cancer. Some tumors, when surgically removed and studied have been found to have both infiltrates of T lymphocytes and antibodies bound to the tumor cells. These antibodies (and other specific immune responses) are assumed to be formed at later stages of the tumor growth, however, even in those cases, serum antibodies have not been reported (probably due to them being mostly "absorbed" by the tumor mass).

Since the mutations of a normal cell that lead to a malignant cell mass involves changes in the structure and function of the cells, it could be assumed that the immune system has recognized some of these changes as antigenic determinants that should be responded against; if so, than the suppression caused by the tumor would be the reason for the lack of antibodies.

If this immune suppression could be overcome, in vitro, it could lead to the formation of antibodies that are not detectable in the serum (we call this process Cimmunology). Identifying the structures that the antibodies bind to, and looking for a correlation between the tumor pathology and the antibodies' specificity - could provide additional information about the tumor - via a blood test.

Future CAAb Test

The Cimmunology based test is comprised of an in-vitro stimulation step and an antibody detection step.

The assay will be used to find Cancer Associated Antibodies in ovarian cancer patients.

Identification of ovarian cancer associated antibodies could provide the clinician with additional immunological and antigenic information regarding the patient's condition or medical status.

The Cimmunology process is comprised of a blood collection and processing step and an incubation (in a special stimulation "tube" called CimTube) period in a humid, 37oC incubator with 5% CO2.

The test for the detection of specific antibodies is ELISA based, and includes different potentially interesting antigens.

The relevant medical and pathological information, to be collected from the patient's file, will enable a more detailed analysis of the test results.

STUDY OBJECTIVES

Primary objective:

* To find Cancer Associated Antibodies

Effectiveness:

* To determine the ability of the Cimmunology process to lead to in vitro antibody production, the ability of the ELISA assays to detect any of those antibodies, and to establish the relationship between the ELISA results and the clinical/pathological status of the patient. The statistical significance of the CAAb test results will be determined.

STUDY POPULATIONS AND PATIENT SELECTION

Ovarian cancer patients

The study population will include subjects that are suspected and going to be treated for ovarian cancer, prior to any surgical procedure or any other anti-cancer treatment. The clinical suspicion includes one of the following: Pelvic mass (by pelvic examination or other imaging techniques), or high CA-125 levels in post menopausal women, ascites, or due to incidental finding of distant metastasis. Final analysis will be done in relation to pathology only.

Control group

The control group will include patients, at the gynecology department (or any other appropriate care unit), with no prior cancer history.

STUDY DESIGN

Overall Description

The current study is a comparative observational two-arm study, involving all consecutive ovarian cancer patients during the study duration, and age matched control subjects. The purpose of the study is to assess the effectiveness of the CAAb test in detecting ovarian cancer associated antibodies.

Subjects will be screened for potential participation in the study, according to the inclusion and exclusion criteria. Patients recruited will be asked to sign an informed consent form.

The data on the patients will include parameters of the clinical and pathological state of the patients, results of CimTube culture step and the experimental kits. The effectiveness of the CAAb test will be assessed by evaluating the statistical significance of the CAAb test used.

The study will utilize a three step group-sequential design with two interim and one final analysis using the O'Brian-Fleming' boundaries. The data collection may be stopped after the first or second interim analysis if the bounds are reached. This could substantially decrease the number of patients and the time of the study, while just slightly increasing the maximum number of patients. (See Sample size considerations below).

We will use 1:2 ratio between cancer and control patients to decrease the necessary number of cancer patients which is the main limiting factor.

The sponsor will conduct an interim analysis, following the first third and second third of ovarian cancer cases and the sample size will be recalculated according to the obtained estimates of the mean and variance of the test in the two groups.

Since the data gathered to date was from epithelial cell carcinoma only, our study will also focus on epithelial cell carcinoma. Therefore stromal and germ cell tumors, which comprise less than 10% of OC cases will be dropped based on the final pathology analysis. In addition, non ovarian cases that were mistaken for ovarian carcinoma comprise approximately 10% of women undergoing surgery for OC. These will also be dropped based on the final pathology.

Therefore, at least 60 patients will be enrolled in the study, in order to obtain the statistically projected needed sample size of 50 ovarian cancer samples. The control group will be 120 patients.

Study Procedure

In the hospital:

First, an identified study patient has to sign an informed consent form, and her Eligibility Form filled; both should be bar-coded.

Patient demographic and clinical information acquired from the patient's medical file, including age, country of origin, medical history and results of tests done leading to the diagnostic evaluation of ovarian cancer (not relevant in the control group) will be recorded on the appropriate, bar-coded, pre-study case report forms. The reports will be either electronic (a dedicated and secured internet site) or via a hard copy. A hard copy of the records will be kept in the department. The study is anonymous and the Department will keep the name of the patient without revealing it to investigators and to the study sponsor.

The Study Sponsor will provide the tubes and the barcode labels for monitoring. The doctor/nurse/phlebotomist will collect three heparin vacuum tubes (20-24 ml), label (bar-code) them, and fill up the initial step in the "Sample follow-up form" (SFF). The tubes with the blood will be packaged in a double sealed container (will be provided by the sponsor). The department will notify the designated shipper to collect the blood up to 1 hour from the time that it has been sampled.

For each OC sample two age matched controls (+/- 3 years) will be recruited too.

Transportation from the Hospital to the Handling Lab:

The blood will be transported at room temperature (18-250C), according to the relevant regulations, to the laboratory. Transportation time will be not more than 6 hours. Times to be recorded in SFF.

In the blood handling laboratory:

The blood handling laboratory (to be located no further than 200km from the collection site) will isolate PBMC (Peripheral blood mononuclear cells) and put them into Cimmunology culture within 20 hours from the sampling time (fill up time in SFF).

The detailed protocol and the Cimmunology media will be provided by Lab Discoveries to the participating laboratories (where applicable). All hospitals in Israel will send the blood samples to the laboratory at Lab Discoveries. After the culture step, the culture fluid will be collected and frozen at -80, in properly labeled aliquots. The frozen samples will be sent to the diagnostic laboratory for antibody tests.

In the diagnostic laboratory:

Antibody tests, such as ELISA, will be prepared using different antigens. The samples will be tested for response to the two antigens that have been identified in the past, and for additional new ones. All the data will be permanently recorded directly into a dedicated computer. For each sample all antibody results will be put into the coded patient file. The results will be analyzed by a statistician with expertise in cancer population studies.

At the Hospital, post surgery:

2-3 weeks after the surgery, the CRO will collect from the patient's file the results from the pathology lab and any other relevant information as to the nature and state of the tumor that was removed during surgery. These results will be recorded on the dedicated and secured internet site and a printed bar-coded CRF-OC will be kept in the Department.

STATISTICAL CONSIDERATIONS

The present study is a comparative observational two-arm study, involving all consecutive ovarian cancer patients during the study duration, and age matched control subjects. The main purpose of the study is to assess the effectiveness of the CAAb tests. This effectiveness will be measured by the Fisher' distance (often called "effect size") d defined as d = |m1-m2|/2 Where m1 is the mean value of the test in the controls, m2 is the mean value in the ovarian cancer patients, |m1-m2| denotes the absolute value of the difference (m1-m2), and s is the common estimate of the standard deviation of the distribution of the test in one group (control or ovarian cancer).

Statistical Hypothesis

Null Hypothesis: There is no relationship between the presence or absence of OC and the CAAb i.e. d=0

Alternative Hypothesis: The expectation of the CAAb in the cancer population differs from that of the control population, i.e. m1 is not equal to m2. Since the sign of the difference is not important, the test will be two-sided.

General Considerations

According to our previous results, we assume that

1. The distributions of the test results in each group are close to Normal or may be transformed to the Normal by log-transformation.
2. The variance of the distributions in the two groups are approximately equal
3. Having in mind that this is a pilot study we will consider the results as significant if the two-sided p-value is 0.1 or less. The bound 0.1 instead of 0.05 was chosen to decrease the chances of random exclusion of some potentially informative tests.

When deciding the continuation of the study no correction for multiple comparisons is assumed. However, the results will be presented without and with the correction using the FDR of Benjamini & Hochberg approach (Benjamini, Hochberg 1995).

Where confidence limits are appropriate, the confidence level will be 95% .

Sample Size

The sample size was calculated using relevant information from our previous study on Peptides P3 and P1 and ovarian cancer. There is no information in the literature regarding cancer associated antibodies.

The sample size is calculated for a three step sequential group design with two sided significance 0.1 and 0.05, power 0.8, for cancer: control ratio 1:2, for D of 0.5. The calculations used the standard formulas for sample size necessary for comparison mean values in two independent groups by t-test. The correction for a group-sequential procedure with O'Bien and Fleming's test increases the numbers by 1.017 and 1.027 for significance values 0.05 and 0.1, that is negligible for our sample sizes. (see C. Jennison, B.W.Turnbill Group Sequential Methods with Applications to Clinical Trials Chapmann & Hall (2000) Boca Raton FL US pp30 table 2.4).

The calculations were done using NCSS-PASS software.

Endpoint Evaluation

Effectiveness Analysis

A calculated D between 0.3 and 0.5 will mark a test as non effective to be used alone. However, it may be important in combination with other tests as a part of the multivariate test procedure. Tests with d < 0.3 will be considered as non-effective. A test, or a combination of tests, with d > 0.5 will mark the CAAb test as effective.

ELIGIBILITY:
Inclusion Criteria:

Ovarian cancer patients:

* Subjects 18 years or over.
* Patients suspected of ovarian cancer (including peritoneal carcinoma). The clinical suspicion will include one of the following: pelvic mass (by pelvic examination or other imaging techniques), or high cancer antigen (CA)-125 levels in post-menopausal women, ascites, or due to incidental finding of distant metastasis. Final analysis will be done in relation to pathology only.
* Patients willing to participate as evidenced by signing the written informed consent.

Control subjects:

* Subjects 18 years or over
* Patients willing to participate as evidenced by signing the written informed consent

Exclusion Criteria:

Ovarian cancer patients:

* Subjects less than 18 years of age
* Hematological malignancies
* Previous ovarian tumor
* Patients under active chemotherapy treatment
* Patients not willing to sign written informed consent

Control subjects:

* Subjects less than 18 years
* Hematological malignancies
* History of any past tumors
* Other ovarian pathology
* Patients who have been under anesthesia in the last 2 months
* Patients treated with immunosuppressant drugs
* Patients not willing to sign written informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2006-07; Study Completion 2008-06

CONTACTS AND LOCATIONS:
Overall Officials: Tamar J. Cohen, Ph.D, Principal Investigator — Lab Discoveries Ltd.
Locations (5):
- Israel (5):
  - Shiba Hospital, Tel Litwinsky, Tel Aviv
  - Soroka, Beersheba
  - Carmel Hospital, Haifa
  - Hadassah Hospital, Ein Karem Campus, Jerusalem
  - Hadassah Hospital, Mt. Scopus Campus, Jerusalem